CLINICAL TRIAL: NCT04778904
Title: A Phase 1b/2a, Open-Label Study to Evaluate the Safety, Tolerability and Immunogenicity of VTP-300 With or Without Nivolumab in Participants With Chronic Hepatitis B Infection
Brief Title: First-In-Human Study of ChAdOx1-HBV & MVA-HBV Vaccines (VTP-300) for Chronic HBV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBV-002; 2020-000190-25 (EudraCT Number)
Record Dates: First submitted 2021-02-01; First posted 2021-03-03 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Nivolumab; Solutions

STUDY DESIGN:
Intervention Model Description: Participants are randomised to the four treatment groups, as the groups are initiated. Allocation to the groups is 1:1:1:1. Version 6.0 of the study protocol has closed Groups 1 and 4 to further randomisation; recruitment will now be in a 1:1 ratio between Groups 2 and 3 only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (MVA-HBV) (Experimental): Day 0: MVA-HBV 1 x 10^8 pfu IM injection Day 28: MVA-HBV 1 x 10^8 pfu IM injection
  Interventions: Biological: MVA-HBV
- Group 2 (ChAdOx1-HBV, MVA-HBV) (Experimental): Day 0: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection Day 28: MVA-HBV 1 x 10^8 pfu IM injection
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV
- Group 3 (ChAdOx1-HBV, MVA-HBV and nivolumab) (Experimental): Day 0: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection Day 28: MVA-HBV 1 x 10^8 pfu IM injection + nivolumab 0.3 mg/kg IV infusion
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV; Biological: Nivolumab
- Group 4 (ChAdOx1-HBV and nivolumab, MVA-HBV and nivolumab) (Experimental): Day 0: ChAdOx1-HBV 1 x 2.5 10^10 vp IM injection + nivolumab 0.3 mg/kg IV infusion Day 28: MVA-HBV 1 x 10^8 pfu IM injection + nivolumab 0.3 mg/kg IV infusion
  Interventions: Biological: ChAdOx1-HBV; Biological: MVA-HBV; Biological: Nivolumab

INTERVENTIONS:
Biological: ChAdOx1-HBV — Chimpanzee Adenovirus Oxford 1-vectored Hepatitis B virus vaccine
  Arms: Group 2 (ChAdOx1-HBV, MVA-HBV); Group 3 (ChAdOx1-HBV, MVA-HBV and nivolumab); Group 4 (ChAdOx1-HBV and nivolumab, MVA-HBV and nivolumab)
Biological: MVA-HBV — Modified Vaccinia Ankara-vectored Hepatitis B virus vaccine
Biological: Nivolumab — Human immunoglobulin G4 monoclonal antibody
  Other Names: Opdivo 10mg/ml concentrate for solution for infusion
  Arms: Group 3 (ChAdOx1-HBV, MVA-HBV and nivolumab); Group 4 (ChAdOx1-HBV and nivolumab, MVA-HBV and nivolumab)

SUMMARY:
This is an open-label study to determine the safety, tolerability and immunogenicity of ChAdOx1-HBV and MVA-HBV vaccines, with or without nivolumab, in patients with chronic HBV who are virally suppressed with oral anti-viral therapies.

DETAILED DESCRIPTION:
This is a multi-centre study conducted in 52 participants, who will each be administered 2 vaccine injections (IM) on Day 0 and Day 28 as follows:

Group 1: MVA-HBV + MVA-HBV (now closed) Group 2: ChAdOx1-HBV + MVA-HBV Group 3: ChAdOx1-HBV + MVA-HBV + nivolumab (IV infusion) Group 4: ChAdOx1-HBV + nivolumab + MVA-HBV + nivolumab (now closed)

Participants are randomised to treatment as the groups are initiated with a 1:1:1:1 allocation. Version 6.0 of the study protocol has closed Groups 1 and 4 to further randomisation; recruitment will now be in a 1:1 ratio between Groups 2 and 3 only. A sentinel participant is dosed in Group 1, with further participants in Group 1 only being dosed at least 48h later. Group 2 is initiated following a Day 7 safety assessment of the first 6 participants in Group 1. Groups 3 and 4 are initiated following a Day 7 safety assessment of the first 6 participants in Group 2.

The primary objective of the study is to determine the safety and reactogenicity of the treatment regimens; this will be assessed by analysis of the incidence and severity of (serious) adverse events and any changes in laboratory values and vital signs.

The secondary objectives of the study are the determination of the immunogenicity of the ChAdOx1-HBV and MVA-HBV vaccines and the impact of PD-blockade, as well as the effect on HBV markers; these are assessed by measurements of the magnitude and avidity of HBV-specific CD4+ and CD8+ T cells and the magnitude of HBV markers.

Following first vaccination, participants remain in the study for 9 months and attend clinic visits for vaccination and assessments on Days 0, 7, 28, 35 and Months, 3, 6 and 9.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged ≥18 to ≤65 years at screening (according to country/local regulations)
2. BMI ≤32kg/m2
3. Able to provide informed consent indicating they understand the purpose of, and procedures required, for the study and are willing to participate
4. If female, willing not to become pregnant up to 8 weeks after last dose of study vaccine and up to 5 months after the last dose of nivolumab
5. If female: Not pregnant or breast feeding and one of the following:

   * Of non-childbearing potential (i.e. women who have had a hysterectomy or tubal ligation or are post menopausal, as defined by no menses in ≥1 year and without an alternative medical cause)
   * Of childbearing potential but agrees to practice highly effective contraception for 4 weeks prior to study vaccine and 8 weeks after study vaccine and 5 months after the last dose of nivolumab. Highly effective methods of contraception include one or more of the following:

     (i) Male partner who is sterile (medically effective vasectomy) prior to the female participant's entry into the study and is the sole sexual partner for the female participant

   (ii) Combined (oestrogen and progestogen-containing) hormonal contraception associated with inhibition of ovulation:
   * oral
   * intravaginal
   * transdermal

   (iii) Progestogen-only hormonal contraception associated with inhibition of ovulation:
   * oral
   * injectable
   * implantable

   (iv) An intrauterine device

   (v) Bilateral tubal occlusion
6. Documented evidence of chronic HBV infection (e.g. HBsAg positive ≥6 months with detectable HBsAg levels at screening)
7. Receipt of only either entecavir, tenofovir (tenofovir alafenamide fumarate or tenofovir disoproxil fumarate), or besifovir for at least 12 months before screening
8. Virally suppressed (HBV-DNA viral load < 40 IU/mL for ≥ 1 year)
9. HBsAg levels <4000 IU/mL

Exclusion Criteria:

1. Presence of any significant acute or chronic, uncontrolled medical/psychiatric illness
2. Hepatitis C virus (HCV) antibody positive.
3. HIV antibody positive
4. Co-infection with hepatitis D virus
5. Documented cirrhosis or advanced fibrosis indicated by a liver biopsy within 6 months prior to screening (Metavir activity grade A3 and stages F3 and F4; Ishak stages 4-6).

   In the absence of a documented liver biopsy, either 1 of the following (not both):
   * Screening Fibroscan with a result > 9 kilopascals (kPa) (or the equivalent) within ≤ 6 months of screening, OR
   * Screening FibroTest >0.48 and aspartate aminotransferase (AST) to platelet ratio index (APRI) of >1.
6. ALT >3 x upper limit of normal (ULN), international normalized ratio (INR) >1.5 unless the participant was stable on an anticoagulant regimen affecting INR, albumin <3.5 g/dL, direct bilirubin >1.5 x ULN, platelet count < 100,000/microlitre.
7. A history of liver decompensation (e.g. ascites, encephalopathy or variceal haemorrhage)
8. Prior hepatocellular carcinoma
9. Chronic liver disease of a non-HBV aetiology
10. History or evidence of autoimmune disease or known immunodeficiency of any cause
11. Presence of active infection
12. Evidence of interstitial lung disease, active pneumonitis, myocarditis, or a history of myocarditis
13. Past history of thyroid disorder or abnormal thyroid function at screening that is still active and uncontrolled
14. Prolonged therapy with immunomodulators (e.g. corticosteroids such as prednisone > 10 mg/day) or biologics (e.g. monoclonal antibodies, IFN) within 3 months of screening
15. Receipt of immunoglobulin or other blood products within 3 months prior to enrolment
16. Receipt of any investigational drug or vaccine within 3 months prior to screening
17. Receipt of any adenoviral-based vaccine within 3 months prior to administration of ChAdOx1-HBV on Day 0, or plan to receive an adenoviral-based vaccine within 3 months after Day 0
18. Receipt of any live vaccines within 30 days prior to screening
19. Receipt of any inactivated vaccines within 14 days prior to screening,
20. History of severe hypersensitivity or anaphylactic reactions likely to be exacerbated by any component of the vaccine or nivolumab
21. Malignancy within 5 years prior to screening with the exception of specific cancers that are cured by surgical resection (e.g. except basal cell skin carcinoma of the skin and cervical carcinoma). Participants under evaluation for possible malignancy are not eligible
22. Current alcohol or substance abuse judged by the Investigator to potentially interfere with participant safety and compliance
23. Significant cardiac disease or unstable uncontrolled cardiac disease
24. Any laboratory test which is abnormal, and which is deemed by the Investigator to be clinically significant
25. Cytotoxic agents, other anti HBV or traditional herbal medicines which, in the opinion of the Investigator, may have activity against HBV within the previous 6 months prior to randomization
26. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Yonsei University College of Medicine, Seoul
  - Asan Medical Centre, Seoul
  - The Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
- Taiwan (4):
  - Buddhist Tzu Chi Medical Foundation, Dalin, Chia-Yi County
  - E-Da Hospital, Kaohsiung City, Yan-chao District
  - Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham, Notts
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Started | 10 | 18 | 18 | 9
Completed | 9 | 18 | 17 | 9
Not Completed | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set consisted of all participants who were randomised.
  Safety analysis set consisted of all participants who received at least 1 vaccination.
  Per-protocol (PP) analysis set consisted of all participants in the safety analysis set who received the correct trial vaccine and who had no major protocol deviations.
  Immunogenicity analysis set consisted of all participants in the PP set who had available immunogenicity data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab) | Total
Number analyzed (Participants) | 10 | 18 | 18 | 9 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 18 | 18 | 9 | 54
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 7 | 2 | 13
  Male | 9 | 15 | 11 | 7 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 18 | 17 | 8 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 6 | 10 | 4 | 20
  Taiwan | 10 | 11 | 6 | 3 | 30
  United Kingdom | 0 | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Participants With Treatment-Emergent Adverse Events (TEAEs) and ≥Grade 3 Study Vaccine-related Adverse Events Following Study Vaccination
Description: The incidence of TEAEs and and ≥Grade 3 study vaccine-related adverse events will be based on the number and percentage of participants with events and number of events.
  TEAEs are defined as all adverse events occurring after study vaccine administration; they will be further categorised by Seriousness, Severity (i.e. ≥ Grade 3) and Causality.
  Seriousness of the TEAEs is assessed according to the published FDA criteria (2016).
  Severity of the TEAEs will be graded according to the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adults and Volunteers Enrolled in Preventative Vaccine Trials, 2007 (70 FR 22664).
Time Frame: From each study vaccination for the following 27 days
Population: Safety analysis set - all participants who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Incidence of vaccine related adverse events following vaccination: Participants experiencing events | 1 | 1 | 2 | 1
  Incidence of vaccine related adverse events following vaccination: No events | 9 | 17 | 16 | 8
  Grade 3 or greater vaccine related adverse events following vaccination: Participants experiencing events | 0 | 0 | 0 | 0
  Grade 3 or greater vaccine related adverse events following vaccination: No events | 10 | 18 | 18 | 9
  Serious Adverse Events vaccine related following vaccination: Participants experiencing events | 0 | 0 | 0 | 0
  Serious Adverse Events vaccine related following vaccination: No events | 10 | 18 | 18 | 9

2. Primary Outcome: The Incidence of Participants With ≥Grade 3 Adverse Events Following Study Vaccination With Nivolumab
Description: The incidence of ≥Grade 3 adverse events will be based on the number and percentage of participants with events and number of events.
  TEAEs are defined as all adverse events occurring after study vaccine administration with nivolumab; they are further categorised by Seriousness, Severity (i.e. ≥ Grade 3) according to FDA Guidance 70 FR 22664 and Causality.
Time Frame: From each study vaccination with nivolumab for the following 27 days
Population: All participants who received at least one vaccination and nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Participants experiencing events | 0 | 0 | 1 | 0
  No events | 10 | 18 | 17 | 9

3. Primary Outcome: The Incidence of Participants With Adverse Events of Special Interest (AESIs)
Description: The incidence of AESIs will be based on the number and percentage of participants with events and number of events.
  AESIs specific to this study include pneumonitis, grade 3 or 4 diarrhoea, diabetes, thyroid diseases, colitis, nephritis, immune-related endocrinopathies, myocarditis, immune-related skin conditions, or other unspecified immune-related adverse reactions.
Time Frame: From study admission (the signature of informed consent) to the end of the study (Month 9)
Population: Safety analysis set - all participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Participants with Adverse Events of Special Interest (AESI) | 0 | 0 | 2 | 0
  Participants with no AESI | 10 | 18 | 16 | 9

4. Primary Outcome: The Incidence of Participants With Treatment-Emergent Adverse Events (TEAEs) Within Each Study Group
Description: The incidence of TEAEs will be based on the number and proportion of participants with events and number of events and will be calculated for each of the four study groups.
Time Frame: From each study vaccination for the following 27 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Participants experiencing events | 6 | 8 | 11 | 4
  No events | 4 | 10 | 7 | 5

5. Primary Outcome: Incidence of Participants With Potentially Clinically Significant Laboratory Signs Within Each Treatment Group as Assessed by the Investigator
Description: The incidence of participants will be based upon the number and proportion of patients in each treatment group with clinically significant laboratory signs (haematology and biochemistry, including liver function tests) as assessed by the investigator.
  All laboratory signs will be reported in SI units. If any laboratory sign is considered to be clinically significant i.e. outside laboratory normal reference range, the severity of this sign will be assessed according to the FDA Guidance for Industry 70 FR 22664. Absolute change, change from baseline and worst change for each participant will be calculated.
  The incidence of participants with treatment-emergent, clinically significant laboratory signs and laboratory signs of Grade 3-4 severity will be calculated for each treatment group at each time point.
Time Frame: From the first vaccination until Month 9 (end of study)
Population: Safety analysis set - participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Haematology: Clinically Significant | 0 | 0 | 2 | 0
  Haematology: Non Clinically Significant | 10 | 18 | 16 | 9
  Biochemistry: Clinically Significant | 0 | 0 | 1 | 0
  Biochemistry: Non Clinically Significant | 10 | 18 | 17 | 9

6. Primary Outcome: Incidence of Participants With Potentially Clinically Significant Vital Signs Within Each Treatment Group as Assessed by the Investigator
Description: The incidence of participants will be based upon the number and proportion of patients in each treatment group with clinically significant vital signs.
  Vital signs will be considered to be potentially clinically significant if they respectively fall below or above the relevant upper and lower limits.
  The incidence of participants with treatment-emergent, clinically significant vital signs will be calculated for each treatment group at each time point.
Time Frame: From the first vaccination until Month 9 (end of study)
Population: Safety Analysis Set - participants who received at least one vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Pulse Rate: Clinically Significant | 0 | 0 | 1 | 0
  Pulse Rate: Non Clinically Significant | 10 | 18 | 17 | 9
  Blood Pressure: Clinically Significant | 1 | 3 | 3 | 2
  Blood Pressure: Non Clinically Significant | 9 | 15 | 15 | 7
  Temperature: Clinically Significant | 0 | 0 | 0 | 0
  Temperature: Non Clinically Significant | 10 | 18 | 18 | 9

7. Primary Outcome: Number of Participants With Worst Changes From Baseline in Laboratory Hematology Parameters
Description: Hematology laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA).
  For all hematology parameters, changes from baseline of at least two severity grades will be calculated for each timepoint at which the laboratory test is conducted throughout the study.
  The number of participants showing shifts of at least two severity grades (as worst change from baseline for each hematology parameter) will be presented within shift tables.
Time Frame: From baseline till Month 9
Population: Statistical Analysis Plan changed analysis of laboratory results so that shift tables of laboratory results, vital signs, and physical examinations were summarised using the worst post-baseline result overall, rather than by time point as indicated in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  WBC decrease: Participants with at least two severity grades change | 0 | 0 | 1 | 0
  WBC decrease: Participants with no change | 10 | 18 | 17 | 9
  WBC increase: Participants with at least two severity grades change | 0 | 0 | 0 | 1
  WBC increase: Participants with no change | 10 | 18 | 18 | 8
  Eosinophils: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Eosinophils: Participants with no change | 10 | 18 | 18 | 9
  Lymphocytes Decrease: Participants with at least two severity grades change | 0 | 0 | 1 | 0
  Lymphocytes Decrease: Participants with no change | 10 | 18 | 17 | 9
  Neutrophils Decrease: Participants with at least two severity grades change | 1 | 0 | 2 | 1
  Neutrophils Decrease: Participants with no change | 9 | 18 | 16 | 8
  Haemoglobin: Participants with at least two severity grades change | 1 | 0 | 0 | 0
  Haemoglobin: Participants with no change | 9 | 18 | 18 | 9
  Platelets decrease: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Platelets decrease: Participants with no change | 10 | 18 | 18 | 9
  Prothrombin time: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Prothrombin time: Participants with no change | 10 | 18 | 18 | 9

8. Primary Outcome: Number of Participants With Worst Changes From Baseline in Laboratory Biochemistry Parameters
Description: Biochemistry laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA).
  For all biochemistry parameters, changes from baseline of at least two severity grades will be calculated for each timepoint at which the laboratory test is conducted throughout the study.
  The number of participants showing shifts of at least two severity grades (as worst change from baseline for each biochemistry parameter) will be presented within shift tables.
Time Frame: From baseline till Month 9
Population: Statistical analysis Plan has changed the planned analysis so that shift tables of laboratory results were summarised using the worst post-baseline result overall, rather than by time point as indicated in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Alanine Aminotransferase: Participants with at least two severity grades change | 0 | 0 | 2 | 0
  Alanine Aminotransferase: Participants with no change | 10 | 18 | 16 | 9
  Aspartate Aminotransferase: Participants with at least two severity grades change | 0 | 0 | 1 | 0
  Aspartate Aminotransferase: Participants with no change | 10 | 18 | 17 | 9
  Alkaline Phosphatase: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Participants with no change | 10 | 18 | 18 | 9
  Bilirubin Increase: Participants with at least two severity grades change | 0 | 1 | 1 | 1
  Bilirubin Increase: Participants with no change | 10 | 17 | 17 | 8
  Blood Urea Nitrogen: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Participants with no change | 10 | 18 | 18 | 9
  Creatinine: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Creatinine: Participants with no change | 10 | 18 | 18 | 9
  Hypokalemia: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Hypokalemia: Participants with no change | 10 | 18 | 18 | 9
  Hyperkalemia: Participants with at least two severity grades change | 0 | 1 | 0 | 0
  Hyperkalemia: Participants with no change | 10 | 17 | 18 | 9
  Hyponatremia: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Hyponatremia: Participants with no change | 10 | 18 | 18 | 9
  Hypernatremia: Participants with at least two severity grades change | 0 | 1 | 1 | 0
  Hypernatremia: Participants with no change | 10 | 17 | 17 | 9
  Hypoalbuminemia: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Hypoalbuminemia: Participants with no change | 10 | 18 | 18 | 9

9. Primary Outcome: Number of Participants With Worst Changes From Baseline in Vital Signs Parameters (Heart Rate, Systolic Blood Pressure, Diastolic Blood Pressure and Temperature)
Description: Worst change is defined as the lowest and highest post-baseline values for heart rate (bradycardia, tachycardia) and systolic blood pressure (hypotension, hypertension), and as the highest post-baseline values for diastolic blood pressure (hypertension) and temperature (fever).
  For all vital signs measurements, changes from baseline will be calculated for each timepoint at which the vital sign measurement is conducted throughout the study.
  The number of participants showing worst change from baseline for the vital signs parameters overall will be presented within shift tables.
Time Frame: From baseline till Month 9
Population: Statistical Analysis Plan changed planned analysis so that shift tables of laboratory results, vital signs, and physical examinations were summarised using the worst post-baseline result overall, rather than by time point as indicated in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Bradycardia: Participants with at least two severity grades change | 0 | 0 | 0 | 2
  Bradycardia: Participants with no change | 10 | 18 | 18 | 7
  Tachycardia: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Tachycardia: Participants with no change | 10 | 18 | 18 | 9
  Hypotension: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Hypotension: Participants with no change | 10 | 18 | 18 | 9
  Hypertension (Systolic): Participants with at least two severity grades change | 1 | 2 | 1 | 1
  Hypertension (Systolic): Participants with no change | 9 | 16 | 17 | 8
  Hypertension (diastolic): Participants with at least two severity grades change | 2 | 3 | 1 | 1
  Hypertension (diastolic): Participants with no change | 8 | 15 | 17 | 8
  Fever: Participants with at least two severity grades change | 0 | 0 | 0 | 0
  Fever: Participants with no change | 10 | 18 | 18 | 9

10. Secondary Outcome: Frequency of HBV-specific CD4+ and CD8+ T Cells Induced by Each Treatment Regimen
Description: The frequency of HBV-specific CD4+ and CD8+ T cells was determined by stimulating Peripheral Blood Mononuclear Cells (PBMC) with peptide pools corresponding to HBV antigens Core, Polymerase and Surface in an Intracellular Cytokine Staining (ICS) flow cytometry assay. In this assay the percentage of CD4+ or CD8+ expressing cytokines IFNγ, IL-2 or TNFα in response to HBV peptides is measured. Frequencies of antigen-specific cytokine-expressing CD4+ or CD8+ T cells are compared across trial timepoints and treatment groups.
Time Frame: Baseline, Day7, Day28, Day35, Month 3, Month 6, Month 9
Population: Immunogenicity Analysis Set
Measure: Median (95% Confidence Interval); unit: percentage of cells
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 9 | 17 | 17 | 9
percentage of cells
  CD4+ Change from Baseline to Day 7 (Core): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD4+ Change from Baseline to Day 7 (Core) | 0.0034 [-0.0277 to 0.0625] | -0.0131 [-0.0382 to 0.0050] | 0.0050 [-0.0344 to 0.0181] | -0.0016 [-0.0178 to 0.0092]
  CD4+ Change from Baseline to Day 28 (Core): number analyzed (Participants) | 9 | 13 | 15 | 8
  CD4+ Change from Baseline to Day 28 (Core) | -0.0089 [-0.0511 to 0.0294] | 0.0050 [-0.0215 to 0.0338] | -0.0003 [-0.0303 to 0.0081] | -0.0051 [-0.0496 to 0.1999]
  CD4+ Change from Baseline to Day 35 (Core): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD4+ Change from Baseline to Day 35 (Core) | -0.0165 [-0.0551 to 0.0336] | -0.0009 [-0.0081 to 0.0208] | -0.0003 [-0.0294 to 0.0182] | -0.0024 [-0.0602 to 0.0818]
  CD4+ Change from Baseline to Month 3 (Core): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD4+ Change from Baseline to Month 3 (Core) | -0.0099 [-0.0551 to 0.0228] | 0.0058 [-0.0098 to 0.0113] | 0.0051 [-0.0437 to 0.0272] | -0.0142 [-0.0796 to 0.1142]
  CD4+ Change from Baseline to Month 6 (Core): number analyzed (Participants) | 9 | 15 | 14 | 7
  CD4+ Change from Baseline to Month 6 (Core) | 0.0128 [-0.0406 to 0.0312] | -0.0163 [-0.0313 to -0.0017] | -0.0213 [-0.0403 to 0.0066] | 0.0197 [-0.1181 to 0.1317]
  CD4+ Change from Baseline to Month 9 (Core): number analyzed (Participants) | 9 | 13 | 14 | 8
  CD4+ Change from Baseline to Month 9 (Core) | 0.0068 [-0.0247 to 0.0334] | -0.0033 [-0.0174 to 0.0363] | -0.0107 [-0.0262 to 0.0200] | -0.0260 [-0.0378 to 0.0177]
  CD4+ Change from Baseline to Day 7 (Pol 1+2): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD4+ Change from Baseline to Day 7 (Pol 1+2) | 0.0068 [-0.0030 to 0.0315] | -0.0040 [-0.0139 to 0.0000] | 0.0020 [0.0000 to 0.0399] | -0.0162 [-0.1309 to 0.0072]
  CD4+ Change from Baseline to Day 28 (Pol 1+2): number analyzed (Participants) | 9 | 13 | 15 | 8
  CD4+ Change from Baseline to Day 28 (Pol 1+2) | 0.0063 [-0.0030 to 0.0245] | 0.0000 [-0.0097 to 0.0016] | 0.0000 [0.0000 to 0.0077] | -0.0155 [-0.1436 to 0.0193]
  CD4+ Change from Baseline to Day 35 (Pol 1+2): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD4+ Change from Baseline to Day 35 (Pol 1+2) | 0.0046 [-0.0018 to 0.0153] | 0.0025 [-0.0097 to 0.0386] | 0.0000 [0.0000 to 0.0153] | -0.0162 [-0.3456 to 0.0201]
  CD4+ Change from Baseline to Month 3 (Pol 1+2): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD4+ Change from Baseline to Month 3 (Pol 1+2) | 0.0068 [-0.0030 to 0.0463] | 0.0000 [-0.0091 to 0.0178] | 0.0002 [0.0000 to 0.0222] | -0.0149 [-0.1094 to 0.0485]
  CD4+ Change from Baseline to Month 6 (Pol 1+2): number analyzed (Participants) | 8 | 15 | 14 | 8
  CD4+ Change from Baseline to Month 6 (Pol 1+2) | 0.0235 [-0.0008 to 0.0567] | 0.0000 [-0.0097 to 0.0067] | 0.0000 [-0.0118 to 0.0170] | -0.0196 [-0.1050 to 0.0555]
  CD4+ Change from Baseline to Month 9 (Pol 1+2): number analyzed (Participants) | 8 | 14 | 14 | 8
  CD4+ Change from Baseline to Month 9 (Pol 1+2) | 0.0066 [-0.0062 to 0.1149] | -0.0011 [-0.0101 to 0.0147] | 0.0000 [0.0000 to 0.0110] | -0.0155 [-0.1639 to 0.0054]
  CD4+ Change from Baseline to Day 7 (Pol 3+4): number analyzed (Participants) | 5 | 14 | 14 | 7
  CD4+ Change from Baseline to Day 7 (Pol 3+4) | 0.0152 [-0.0838 to 0.0737] | -0.0035 [-0.0436 to 0.0204] | -0.0023 [-0.0166 to 0.0188] | -0.0218 [-0.0579 to 0.0266]
  CD4+ Change from Baseline to Day 28 (Pol 3+4): number analyzed (Participants) | 5 | 13 | 15 | 7
  CD4+ Change from Baseline to Day 28 (Pol 3+4) | -0.0076 [-0.0258 to 0.0827] | 0.0028 [-0.0291 to 0.0191] | 0.0000 [-0.0261 to 0.0126] | -0.0324 [-0.0729 to 0.0493]
  CD4+ Change from Baseline to Day 35 (Pol 3+4): number analyzed (Participants) | 6 | 15 | 14 | 6
  CD4+ Change from Baseline to Day 35 (Pol 3+4) | 0.0052 [-0.1305 to 0.0688] | 0.0093 [-0.0283 to 0.0341] | 0.0000 [-0.0098 to 0.0303] | -0.0191 [-0.0562 to 0.0412]
  CD4+ Change from Baseline to Month 3 (Pol 3+4): number analyzed (Participants) | 5 | 14 | 15 | 7
  CD4+ Change from Baseline to Month 3 (Pol 3+4) | 0.0109 [-0.1014 to 0.0492] | 0.0007 [-0.0098 to 0.0174] | 0.0120 [-0.0257 to 0.0369] | -0.0232 [-0.0869 to 0.1094]
  CD4+ Change from Baseline to Month 6 (Pol 3+4): number analyzed (Participants) | 6 | 14 | 14 | 7
  CD4+ Change from Baseline to Month 6 (Pol 3+4) | 0.0066 [-0.1055 to 0.0395] | 0.0022 [-0.0183 to 0.0653] | -0.0034 [-0.0194 to 0.0575] | -0.0232 [-0.0611 to 0.1405]
  CD4+ Change from Baseline to Month 9 (Pol 3+4): number analyzed (Participants) | 6 | 13 | 14 | 8
  CD4+ Change from Baseline to Month 9 (Pol 3+4) | 0.0058 [-0.0767 to 0.0243] | 0.0069 [-0.0143 to 0.0453] | 0.0154 [-0.0489 to 0.0270] | -0.0267 [-0.0419 to 0.0247]
  CD4+ Change from Baseline to Day 7 (Pre-S1/S2+S): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD4+ Change from Baseline to Day 7 (Pre-S1/S2+S) | 0.0071 [-0.0249 to 0.0441] | -0.0372 [-0.0862 to 0.0177] | -0.0173 [-0.0550 to 0.0163] | -0.0117 [-0.0954 to 0.0300]
  CD4+ Change from Baseline to Day 28 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 13 | 15 | 7
  CD4+ Change from Baseline to Day 28 (Pre-S1/S2+S) | 0.0022 [-0.0484 to 0.0929] | 0.0058 [-0.0203 to 0.0148] | -0.0210 [-0.0679 to 0.0088] | -0.0304 [-0.0627 to 0.0057]
  CD4+ Change from Baseline to Day 35 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD4+ Change from Baseline to Day 35 (Pre-S1/S2+S) | -0.0162 [-0.0727 to 0.0478] | 0.0031 [-0.0318 to 0.0705] | -0.0363 [-0.0639 to 0.0244] | -0.0260 [-0.0724 to 1.3927]
  CD4+ Change from Baseline to Month 3 (Pre-S1/S2+S): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD4+ Change from Baseline to Month 3 (Pre-S1/S2+S) | -0.0166 [-0.0332 to 0.0329] | 0.0005 [-0.0252 to 0.0269] | -0.0319 [-0.0824 to 0.0373] | 0.0158 [-0.1124 to 0.0621]
  CD4+ Change from Baseline to Month 6 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 15 | 14 | 8
  CD4+ Change from Baseline to Month 6 (Pre-S1/S2+S) | 0.0107 [-0.0318 to 0.0575] | -0.0119 [-0.0556 to 0.0393] | -0.0202 [-0.0869 to 0.0428] | -0.0215 [-0.0396 to 0.0866]
  CD4+ Change from Baseline to Month 9 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 14 | 13 | 8
  CD4+ Change from Baseline to Month 9 (Pre-S1/S2+S) | 0.0052 [-0.0188 to 0.0347] | -0.0011 [-0.0384 to 0.0512] | -0.0249 [-0.1262 to 0.0210] | -0.0270 [-0.0364 to 0.0233]
  CD8+ Change from Baseline to Day 7 (Core): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD8+ Change from Baseline to Day 7 (Core) | 0.0027 [-0.0556 to 0.0975] | 0.0000 [-0.0353 to 0.0262] | -0.0010 [-0.0357 to 0.0573] | -0.0231 [-0.0853 to 0.1737]
  CD8+ Change from Baseline to Day 28 (Core): number analyzed (Participants) | 9 | 13 | 15 | 8
  CD8+ Change from Baseline to Day 28 (Core) | 0.0054 [-0.0421 to 0.1203] | 0.0000 [-0.0575 to 0.0098] | -0.0203 [-0.0553 to 0.0245] | -0.0011 [-0.0182 to 0.0412]
  CD8+ Change from Baseline to Day 35 (Core): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD8+ Change from Baseline to Day 35 (Core) | -0.0194 [-0.0442 to 0.0299] | 0.0003 [-0.0078 to 0.0815] | 0.0000 [-0.0455 to 0.0285] | 0.0000 [-0.0496 to 0.1169]
  CD8+ Change from Baseline to Month 3 (Core): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD8+ Change from Baseline to Month 3 (Core) | -0.0364 [-0.1506 to 0.0280] | 0.0147 [-0.0208 to 0.0617] | -0.0204 [-0.0553 to 0.0081] | 0.0008 [-0.0804 to 0.0334]
  CD8+ Change from Baseline to Month 6 (Core): number analyzed (Participants) | 9 | 15 | 14 | 7
  CD8+ Change from Baseline to Month 6 (Core) | 0.0108 [-0.1378 to 0.0819] | 0.0145 [-0.0119 to 0.0578] | -0.0219 [-0.0568 to 0.0097] | -0.0061 [-0.0737 to 0.1041]
  CD8+ Change from Baseline to Month 9 (Core): number analyzed (Participants) | 9 | 13 | 14 | 8
  CD8+ Change from Baseline to Month 9 (Core) | 0.0000 [-0.1506 to 0.0467] | 0.0092 [-0.0033 to 0.0951] | 0.0038 [-0.0215 to 0.0341] | -0.0001 [-0.0440 to 0.0724]
  CD8+ Change from Baseline to Day 7 (Pol 1+2): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD8+ Change from Baseline to Day 7 (Pol 1+2) | 0.0000 [-0.0131 to 0.0662] | 0.0000 [0.0000 to 0.0000] | 0.0000 [-0.0179 to 0.0621] | -0.0018 [-0.1589 to 0.0481]
  CD8+ Change from Baseline to Day 28 (Pol 1+2): number analyzed (Participants) | 9 | 13 | 15 | 8
  CD8+ Change from Baseline to Day 28 (Pol 1+2) | 0.0000 [-0.0131 to 0.0265] | 0.0000 [-0.0286 to 0.0060] | 0.0000 [-0.0004 to 0.0267] | -0.0276 [-0.1589 to 0.0000]
  CD8+ Change from Baseline to Day 35 (Pol 1+2): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD8+ Change from Baseline to Day 35 (Pol 1+2) | 0.0000 [-0.0150 to 0.0000] | 0.0000 [0.0000 to 0.0370] | 0.0010 [-0.0102 to 0.0345] | -0.0401 [-0.7508 to 0.0135]
  CD8+ Change from Baseline to Month 3 (Pol 1+2): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD8+ Change from Baseline to Month 3 (Pol 1+2) | 0.0146 [-0.0150 to 0.1076] | 0.0018 [0.0000 to 0.0446] | 0.0000 [0.0000 to 0.0025] | 0.0000 [-0.1354 to 0.0196]
  CD8+ Change from Baseline to Month 6 (Pol 1+2): number analyzed (Participants) | 8 | 15 | 14 | 8
  CD8+ Change from Baseline to Month 6 (Pol 1+2) | 0.0058 [0.0000 to 0.1146] | 0.0009 [0.0000 to 0.0304] | 0.0000 [-0.0047 to 0.0275] | -0.0085 [-0.1068 to 0.0058]
  CD8+ Change from Baseline to Month 9 (Pol 1+2): number analyzed (Participants) | 8 | 14 | 14 | 8
  CD8+ Change from Baseline to Month 9 (Pol 1+2) | 0.0000 [-0.0075 to 0.0802] | 0.0054 [0.0000 to 0.0404] | 0.0000 [-0.0085 to 0.0288] | -0.0152 [-0.1589 to 0.0044]
  CD8+ Change from Baseline to Day 7 (Pol 3+4): number analyzed (Participants) | 5 | 14 | 14 | 7
  CD8+ Change from Baseline to Day 7 (Pol 3+4) | 0.0189 [-0.0345 to 0.1001] | -0.0055 [-0.0415 to 0.0098] | 0.0322 [-0.0213 to 0.1084] | -0.0443 [-0.1450 to 0.0363]
  CD8+ Change from Baseline to Day 28 (Pol 3+4): number analyzed (Participants) | 5 | 13 | 15 | 7
  CD8+ Change from Baseline to Day 28 (Pol 3+4) | -0.0075 [-0.0523 to 0.1291] | 0.0051 [-0.0271 to 0.0647] | 0.0004 [-0.0358 to 0.0579] | -0.0161 [-0.1284 to 0.0796]
  CD8+ Change from Baseline to Day 35 (Pol 3+4): number analyzed (Participants) | 6 | 15 | 14 | 6
  CD8+ Change from Baseline to Day 35 (Pol 3+4) | -0.0021 [-0.0754 to 0.0883] | 0.0131 [-0.0043 to 0.1186] | 0.0477 [0.0006 to 0.1503] | 0.0144 [-0.2188 to 0.5461]
  CD8+ Change from Baseline to Month 3 (Pol 3+4): number analyzed (Participants) | 5 | 14 | 15 | 7
  CD8+ Change from Baseline to Month 3 (Pol 3+4) | 0.0375 [-0.0235 to 0.0757] | 0.0180 [-0.0228 to 0.2331] | 0.0110 [-0.0318 to 0.0749] | -0.0430 [-0.2208 to 0.1043]
  CD8+ Change from Baseline to Month 6 (Pol 3+4): number analyzed (Participants) | 6 | 14 | 14 | 7
  CD8+ Change from Baseline to Month 6 (Pol 3+4) | 0.0318 [-0.0373 to 0.1127] | 0.0096 [-0.0267 to 0.0980] | 0.0138 [-0.0042 to 0.1727] | -0.0585 [-0.2379 to 0.1120]
  CD8+ Change from Baseline to Month 9 (Pol 3+4): number analyzed (Participants) | 6 | 13 | 14 | 8
  CD8+ Change from Baseline to Month 9 (Pol 3+4) | 0.0478 [-0.0746 to 0.2997] | 0.0068 [-0.0329 to 0.0804] | 0.0412 [-0.0138 to 0.0888] | -0.0634 [-0.0906 to 0.2202]
  CD8+ Change from Baseline to Day 7 (Pre-S1/S2+S): number analyzed (Participants) | 8 | 15 | 14 | 7
  CD8+ Change from Baseline to Day 7 (Pre-S1/S2+S) | 0.0054 [-0.0262 to 0.1085] | 0.0042 [-0.0301 to 0.0525] | -0.0034 [-0.0491 to 0.1314] | -0.0574 [-0.1699 to 0.1008]
  CD8+ Change from Baseline to Day 28 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 13 | 15 | 7
  CD8+ Change from Baseline to Day 28 (Pre-S1/S2+S) | 0.0000 [-0.0774 to 0.0462] | 0.0065 [-0.0871 to 0.0304] | -0.0130 [-0.1008 to 0.0711] | -0.0120 [-0.1582 to 0.0990]
  CD8+ Change from Baseline to Day 35 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 15 | 15 | 7
  CD8+ Change from Baseline to Day 35 (Pre-S1/S2+S) | -0.0093 [-0.2066 to 0.0000] | 0.0000 [-0.0265 to 0.0999] | 0.0000 [-0.0484 to 0.0651] | -0.0446 [-0.1609 to 0.7839]
  CD8+ Change from Baseline to Month 3 (Pre-S1/S2+S): number analyzed (Participants) | 6 | 14 | 15 | 7
  CD8+ Change from Baseline to Month 3 (Pre-S1/S2+S) | -0.0304 [-0.0881 to 0.0524] | 0.0385 [0.0000 to 0.1025] | -0.0292 [-0.0802 to 0.0000] | -0.0390 [-0.2847 to 0.1337]
  CD8+ Change from Baseline to Month 6 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 15 | 14 | 8
  CD8+ Change from Baseline to Month 6 (Pre-S1/S2+S) | 0.0481 [-0.2066 to 0.1186] | 0.0000 [-0.0650 to 0.0267] | 0.0215 [-0.0376 to 0.0713] | -0.0246 [-0.1491 to 0.1077]
  CD8+ Change from Baseline to Month 9 (Pre-S1/S2+S): number analyzed (Participants) | 9 | 14 | 13 | 8
  CD8+ Change from Baseline to Month 9 (Pre-S1/S2+S) | 0.0012 [0.0000 to 0.0897] | 0.0195 [-0.0221 to 0.1407] | -0.0130 [-0.1505 to 0.1012] | 0.0006 [-0.1844 to 0.1839]

11. Secondary Outcome: Percentage of Participants With Reduction in HBsAg Titre
Description: This will be determined from samples of PBMCs. The percentage of participants with a HBsAg loss >0.5 log10 and >1.0 log10 will be determined for each vaccine and for each treatment group.
Time Frame: Baseline, Day7, Day28, Day35, Month 3, Month 6, Month 9
Population: Per Protocol population used for HBsAg changes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Loss from Baseline to Day 7: > 0.5 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 7: > 1.0 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 7: No log change or <0.5 log10 | 10 | 18 | 18 | 9
  Loss from Baseline to Day 28: number analyzed (Participants) | 9 | 17 | 18 | 9
  Loss from Baseline to Day 28: > 0.5 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 28: > 1.0 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 28: No log change or <0.5 log10 | 9 | 17 | 18 | 9
  Loss from Baseline to Day 35: number analyzed (Participants) | 9 | 18 | 18 | 9
  Loss from Baseline to Day 35: > 0.5 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 35: > 1.0 log10 | 0 | 0 | 0 | 0
  Loss from Baseline to Day 35: No log change or <0.5 log10 | 9 | 18 | 18 | 9
  Loss from Baseline to Month 3: number analyzed (Participants) | 9 | 18 | 18 | 9
  Loss from Baseline to Month 3: > 0.5 log10 | 0 | 3 | 7 | 1
  Loss from Baseline to Month 3: > 1.0 log10 | 0 | 1 | 4 | 0
  Loss from Baseline to Month 3: No log change or <0.5 log10 | 9 | 14 | 7 | 8
  Loss from Baseline to Month 6: number analyzed (Participants) | 9 | 18 | 18 | 9
  Loss from Baseline to Month 6: > 0.5 log10 | 1 | 3 | 4 | 0
  Loss from Baseline to Month 6: > 1.0 log10 | 0 | 2 | 4 | 0
  Loss from Baseline to Month 6: No log change or <0.5 log10 | 8 | 13 | 10 | 9
  Loss from Baseline to Month 9: number analyzed (Participants) | 9 | 18 | 17 | 9
  Loss from Baseline to Month 9: > 0.5 log10 | 1 | 3 | 5 | 0
  Loss from Baseline to Month 9: > 1.0 log10 | 0 | 1 | 4 | 0
  Loss from Baseline to Month 9: No log change or <0.5 log10 | 8 | 14 | 8 | 9

12. Secondary Outcome: Percentage of Participants With HBsAg and HBeAg Loss
Description: The proportion of participants infected with HBsAg-positive virus at baseline who develop Hepatitis B surface antigen antibody will be determined for each vaccine and for each treatment group.
  The proportion of participants infected with HBeAg-positive virus at baseline who develop Hepatitis B e-antigen antibody will be determined for each vaccine and for each treatment group.
Time Frame: Baseline, Month 9
Population: Intent to Treat Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  HBsAg Seroconversion at Month 9: number analyzed (Participants) | 9 | 18 | 17 | 9
  HBsAg Seroconversion at Month 9: Seroconversion | 0 | 0 | 2 | 0
  HBsAg Seroconversion at Month 9: No Seroconversion | 9 | 18 | 15 | 9
  HBeAg Seroconversion1 at Month 9: number analyzed (Participants) | 1 | 4 | 5 | 3
  HBeAg Seroconversion1 at Month 9: Seroconversion | 0 | 1 | 2 | 1
  HBeAg Seroconversion1 at Month 9: No Seroconversion | 1 | 3 | 3 | 2

13. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: The proportion of participants infected with HBsAg-positive virus at baseline who become HBsAg negative will be determined for each vaccine and for each treatment group.
  The times to seroconversion will be calculated in months.
Time Frame: Baseline and Month 9
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 9 | 18 | 17 | 9
Participants
  No seroconversion (i.e., HBsAg > LLoQ) at Month 9 | 9 | 18 | 15 | 9
  Seroconversion (i.e., HBsAg < LLoQ) at Month 9 | 0 | 0 | 2 | 0

14. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion
Description: This will be determined from samples of PBMCs. The proportion of participants infected with HBeAg-positive virus at baseline who become HBeAg negative will be determined for each vaccine and for each treatment group.
  The times to seroconversion will be calculated in months.
Time Frame: Baseline and Month 9
Population: ITT Analysis Set The overall number of particpants analyized is made up of number of participants who are HBeAg positive at baseline and have non-missing HBeAg results at Month 9. This results in a smaller analysis population than the total participants for each group
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 1 | 4 | 5 | 3
Participants
  Seroconversion | 0 | 1 | 2 | 1
  No Seroconversion | 1 | 3 | 3 | 2

15. Secondary Outcome: Percentage of Participants With Reduction of Hepatitis B DNA
Description: Changes from baseline will be calculated for each vaccine and for each treatment group.
Time Frame: Baseline, Day 35, Month 3 and Month 9
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
Number analyzed (Participants) | 10 | 18 | 18 | 9
Participants
  Baseline: No HBV DNA detected | 7 | 16 | 14 | 7
  Baseline: < 20 IU/mL HBV DNA detected | 3 | 2 | 4 | 2
  Baseline: ≥ 20 IU/mL HBV DNA detected | 0 | 0 | 0 | 0
  Day 35: number analyzed (Participants) | 9 | 18 | 18 | 9
  Day 35: No HBV DNA detected | 8 | 10 | 10 | 8
  Day 35: < 20 IU/mL HBV DNA detected | 1 | 7 | 6 | 1
  Day 35: ≥ 20 IU/mL HBV DNA detected | 0 | 1 | 2 | 0
  Month 3: number analyzed (Participants) | 9 | 18 | 18 | 9
  Month 3: No HBV DNA detected | 6 | 14 | 13 | 7
  Month 3: < 20 IU/mL HBV DNA detected | 3 | 4 | 5 | 2
  Month 3: ≥ 20 IU/mL HBV DNA detected | 0 | 0 | 0 | 0
  Month 9: number analyzed (Participants) | 10 | 18 | 17 | 9
  Month 9: No HBV DNA detected | 10 | 16 | 16 | 7
  Month 9: < 20 IU/mL HBV DNA detected | 0 | 2 | 1 | 2
  Month 9: ≥ 20 IU/mL HBV DNA detected | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of Informed Consent signature by participants (up to 1.5 months prior to first dose) to End of Study (9 months from first dose), that is up 10.5 months
Description: Adverse Events were recorded in the eCRF from the date the informed consent is signed, at all clinic visits to cover the period since the previous visit and during the visit.
  Serious adverse events and adverse events of special interest were recorded from the date the informed consent is signed until the end of the study or resolved or until participant contact discontinues
Arm/Group | Group 1 (MVA-HBV) | Group 2 (ChAdOx1-HBV, MVA-HBV) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18 | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/18 | 1/18 | 0/9
Other Adverse Events (participants affected / at risk) | 6/10 | 8/18 | 11/18 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (MVA-HBV) (N=10) | Group 2 (ChAdOx1-HBV, MVA-HBV) (N=18) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) (N=18) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab) (N=9)
RHEGMATOGENOUS RETINAL DETACHMENT OD (RIGHT EYE (OCULUS DEXTER) (Eye disorders) | 1 (1) | NA | 0 (0) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | NA | 1 (1) | NA
POLYPOSIS OVER RIGHT MAXILARY SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | NA | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (MVA-HBV) (N=10) | Group 2 (ChAdOx1-HBV, MVA-HBV) (N=18) | Group 3 (ChAdOx1-HBV, MVA-HBV and Nivolumab) (N=18) | Group 4 (ChAdOx1-HBV and Nivolumab, MVA-HBV and Nivolumab) (N=9)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal metaplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement restricting the right of the Participating Organisation and/or Principal Investigator to publish trial results, which may not be before the first multi-site publication. Following this, Participating Organisation and/or Principal Investigator may publish results, subject to Sponsor's prior review and comment (within 60 days). Sponsor can request a delay of publication up to six (6) months to enable protection of its proprietary information and/or IPR and know-how.

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT04778904/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04778904/SAP_001.pdf